CLINICAL TRIAL: NCT04070586
Title: ADAPT: Adaptive CT Acquisition for Personalised Thoracic Imaging: A Phase 1 Pilot Study on the Use of Respiratory Motion Guided 4DCBCT for Lung Cancer Radiotherapy
Brief Title: Adaptive CT Acquisition for Personalised Thoracic Imaging
Acronym: ADAPT
Status: Completed | Type: Observational
Sponsor: University of Sydney (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Liverpool Cancer Therapy Centre (Other Government)
Responsible Party: Sponsor
Other Study IDs: HREC/18/LPOOL/361
Record Dates: First submitted 2019-08-13; First posted 2019-08-28 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Cancer, Lung
Keywords: Lung cancer; Radiotherapy; 4DCBCT
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 4DCBCT images: 4DCBCT images are acquired and assessed offline.
  Interventions: Device: 4DCBCT images

INTERVENTIONS:
Device: 4DCBCT images — Images are acquired and assessed offline

SUMMARY:
In this trial, Respiratory Motion Guided (RMG) 4DCBCT will be implemented for the first time on lung cancer patients. RMG-4DCBCT adapts the image acquisition as the patient's breathing changes (i.e. if the patient breathes faster, imaging data is acquired faster).

By adapting the acquisition to the dynamic patient, personalised images of a patients lungs are able to be acquired for radiotherapy treatments.

DETAILED DESCRIPTION:
Four dimensional cone beam computed tomography (4DCBCT) continues to play a pivotal role in the safe delivery of radiotherapy treatments for lung cancer patients. 4DCBCT meets exacting tumour localisation requirements by allowing radiation therapists to measure the tumour as a patient breathes (4D=volumetric images plus respiratory induced tumour motion). Despite the success of 4DCBCT to date, it suffers from relatively poor image quality, very long scan times (4min) and higher imaging doses than are necessary. The primary reason for these problems is that although the purpose of 4DCBCT is to acquire information about tumour motion due to respiration, there is no feedback from the patients breathing signal to adapt and optimise the image acquisition process. This clinical trial is a phase 1 first in human's pilot study and the aim is therefore to prove feasibility of RMG-4DCBCT, not necessarily efficacy. As such, patient scans will be acquired across a broad range of patient breathing conditions to optimise the RMG-4DCBCT technique and also to plan a hypothesis driven clinical trial to follow.

ELIGIBILITY:
Inclusion Criteria:

* Have the ability to give informed consent
* A diagnosis of lung cancer with an indication for radiotherapy either curative or palliative
* Radiotherapy treatment involving the routine acquisition of CBCT for patient setup provided that 4DCBCT is to be acquired during the course of treatment.
* At least two radiotherapy fractions during the course of treatment.

Exclusion Criteria:

* Pregnant women.
* Patient who in the opinion of the treating physician could not tolerate the extra time on the treatment couch for two days of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung cancer who will be treated with radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
RMG-4DCBCT image guidance is feasible for lung cancer patients undergoing radiotherapy | 2 years
  This will be achieved by performing (offline) analysis of the RMG-4DCBCT images obtained and scoring them on a scale of one (excellent quality for image guidance) to three (unsuitable for image guidance).

SECONDARY OUTCOMES:
To measure the extent of association between image quality and the patients' breathing conditions. | 2 years
  Using RMG-4DCBCT scans acquired across a broad range of patients for the first time we will determine if there is a link between image quality and the patients' breathing conditions. This information will be used to improve the prototype.

CONTACTS AND LOCATIONS:
Overall Officials: Ricky O'Brien, PhD, Principal Investigator — University of Sydney
Locations (1):
- Liverpool Hospital, Liverpool, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Only non-identifiable data may be made available for other scientific research, e.g., nonidentifiable data placed on a well-controlled university site, upon request. The data sharing platform is a secure on-line storage solution ("CloudStor") provided through University of Sydney. The data will be stored as a password-protected, encrypted file. In order to download or decompress the data, participating researchers agree to the terms of use for the data, including: (i) that the data is not to be published or otherwise redistributed without the express consent of the original investigators.
Supporting Information: Study Protocol
Time Frame: Data will become available following completion of the final analysis. Data will be available indefinitely.
Access Criteria: Data will be made available to other researchers upon request.

REFERENCES:
- [Derived] Lau BKF, Reynolds T, Keall PJ, Sonke JJ, Vinod SK, Dillon O, O'Brien RT. Reducing 4DCBCT imaging dose and time: exploring the limits of adaptive acquisition and motion compensated reconstruction. Phys Med Biol. 2022 Mar 7;67(6). doi: 10.1088/1361-6560/ac55a4. PMID 35172286